CLINICAL TRIAL: NCT07346911
Title: Digital Interventions for Relapse Prevention in Adolescence
Acronym: DigiTIFF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Ragnhild Bø, Researcher, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 870757
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Major Depression Disorder; ANXIETY DISORDERS (or Anxiety and Phobic Neuroses)
Keywords: Transdiagnostic interventions
MeSH Terms: conditions — Anxiety Disorders; Phobic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App intervention (Experimental): A transdiagnostic, self-guided CBT app:
  1. Standardized self-assessment for mental health: 'Test your psychological immune system'.
  2. Educational mini-series: A 30-minute, entertaining video series that teaches users to build resilience by addressing essential needs like sleep (psychological immune system), recognizing negative thought patterns (thought viruses), and developing healthier coping mechanisms (psychological vitamins).
  3. Daily practice: Over 20 days, users receive a short, 1-2-minute video each morning. These videos provide practical tips, small experiments, or simple tasks designed to help users integrate healthier coping strategies into their daily lives.
  Interventions: Behavioral: Transdiagnostic app intervention
- Group intervention (Experimental): A transdiagnostic, mastery course for groups, delivered weekly in webinar format over three sessions. It includes videos and group discussions.
  Interventions: Behavioral: Transdiagnostic mastery course
- Assessment only (No Intervention): Only assessment will be conducted.

INTERVENTIONS:
Behavioral: Transdiagnostic app intervention — A transdiagnostic, self-guided CBT app, called TankeVirus (literally translated Thought Viruses), consisting of three components:
  1. Standardized self-assessment for mental health: 'Test your psychological immune system'.
  2. Educational mini-series: A 30-minute, entertaining video series that teaches users to build resilience by addressing essential needs like sleep (psychological immune system), recognizing negative thought patterns (thought viruses), and developing healthier coping mechanisms (psychological vitamins).
  3. Daily practice: Over 20 days, users receive a short, 1-2-minute video each morning. These videos provide practical tips, small experiments, or simple tasks designed to help users integrate healthier coping strategies into their daily lives.
  Arms: App intervention
Behavioral: Transdiagnostic mastery course — Group-based webinar offering psychoeducation based on principles of CBT.
  Arms: Group intervention

SUMMARY:
Some adolescents experience periods of anxiety and/or depression, and some find that these periods return over time. The purpose of this study is to examine whether digital interventions-where individuals work systematically with their own thoughts and feelings during periods when they feel well-can help them maintain well-being for longer.

The study includes adolescents aged 16-19 who have previously experienced episodes of depression and/or anxiety to a degree that led them to seek help (e.g., from a school nurse, general practitioner, health clinic, or child and adolescent mental health service). Through a research app on their smartphones, participants complete tasks and answer questionnaires. The study is fully digital. Some participants meet with a therapist in digital group sessions, while others work independently with the digital content.

We will also examine the cost-benefit aspects of offering such interventions. If the study achieves its goals, digital interventions may eventually become a service offered to adolescents recovering from depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Currently in full or partial remission for a minimum of 2 months from a depressive disorder or an anxiety disorder.
* Native or fluent Scandinavian language skills.
* Willingness to take part even when allocated to the non-preferred arm of the trial.

Exclusion Criteria:

* Ongoing depressive disorder, ongoing anxiety disorder.
* Recent completion of one of the interventions in the two interventional arms.
* no available smartphone.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 495 (Estimated)
Dates: Start 2026-04-07 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Relapse: Number of participants scoring above the diagnostic cut-off on the PHQ-9 modified for teens during the 12-month follow-up. | From enrollment to the end of follow-up at 12-months.
  To use the PHQ-9 as a diagnostic aid for Major Depressive Disorder:
  * Questions 1 and/or 2 need to be endorsed as a "2" or "3"
  * Need five or more positive symptoms (positive is defined by a "2" or "3" in questions 1-8 and "1", "2", or "3" in question 9).
  * The functional impairment question (How difficult….) needs to be rated at least as "somewhat difficult."
Time until relapse; reaching the diagnostic criteria of MDD according to PHQ-9 modified for teens | From enrollment to 12-months follow-up
  Number of days until the diagnostic criteria of MDD as assessed PHQ-9 modified for teens has been reached.
  - Questions 1 and/or 2 need to be endorsed as a "2" or "3"
  * Need five or more positive symptoms (positive is defined by a "2" or "3" in questions 1-8 and by a "1", "2", or "3" in question 9).
  * The functional impairment question (How difficult….) needs to be rated at least as "somewhat difficult."

SECONDARY OUTCOMES:
Repetitive negative thinking (RNT-10) | At enrollment, and at 3, 6 and 12 months follow-up
  Assess transdiagnostic repetitive negative thinking
Somatic complaints (SSS8) | At enrollment, and at 3, 6, and 12-months follow-up.
  Somatic complaints based on sum score of all items
EPOCH Measure of Adolescent Well-Being | At baseline, 3, 6 and 12-months follow-up.
  A 20-item validated questionnaire (4 items per domain; Engagement, Perseverance, Optimism, Connectedness, Happiness) on a 1-5 Likert scale (1=Almost Never, 5=Almost Always) resulting in domain scores, reflecting strengths in these positive psychological areas crucial for youth well-being.
Health related quality of life | At baseline, 3, 6 and 12-months follow-up.
  EQ-5D-5L will be used to assess five domains of patient reported outcomes and for economic evaluation of the interventions.
Health related quality of life - Visual Analog Scale | At baseline, 3, 6 and 12-months follow-up.
  EQ VAS will be used to assess patient reported outcomes for self-rated health and for economic evaluation of the interventions.

OTHER OUTCOMES:
Client satisfaction questionnaires (CSQ-I) | At 3 months follow-up.
  The 8-item questionnaire assesses how satisfied the participants are with the interventions, only administrated to those who are in the interventional arms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The dataset underlying the results will be shared together with publications.

REFERENCES:
- See also: Project webpage — https://www.sv.uio.no/psi/english/research/projects/digitiff/

DOCUMENTS (1):
  • Study Protocol (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT07346911/Prot_000.pdf